CLINICAL TRIAL: NCT07277413
Title: A Multicenter Study Evaluating the Safety, Efficacy, and Pharmacokinetics of IDE892 as Monotherapy and Combination Therapy in Participants With MTAP-Deleted Advanced Solid Tumors
Brief Title: A Study of IDE892 as Monotherapy and Combination in MTAP-deleted Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: IDEAYA Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDE892-001
Record Dates: First submitted 2025-11-13; First posted 2025-12-11 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: NSCLC Adenocarcinoma; Gastroesophageal Cancer (GC); Gastric Adenocarcinoma; Adenocarcinoma of Esophagus; Squamous Cell Car. - Esophagus; Urothelial Carcinoma (UC); Bladder Cancer; Mesothelioma; Pleural Mesothelioma; Peritoneal Mesothelioma; Non-Small Cell Lung Cancer NSCLC
Keywords: MTAP deletion; MTAP loss; MTAP-deficient tumors; homozygous MTAP loss; IDE892; IDE397; MAT2A inhibitor; PRMT5; advanced solid tumors; metastatic cancer; recurrent cancer; dose escalation; dose expansion; phase 1 clinical trial; ctDNA
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Mesothelioma; Mesothelioma, Malignant; Neoplasm Metastasis; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1: IDE892 Monotherapy Dose Escalation (MTAP-deleted advanced solid tumors) (Experimental): Participants with advanced or metastatic solid tumors harboring MTAP deletion (including mesothelioma, gastroesophageal cancers, non-small cell lung cancer, and urothelial cancer) will receive IDE892. Dose levels will be escalated sequentially using a Bayesian Optimal Interval (BOIN) design to evaluate safety, tolerability, and to determine the maximum tolerated dose and/or recommended dose for expansion. PK and pharmacodynamics (PD) and preliminary antitumor activity will also be assessed.
  Interventions: Drug: IDE892
- Part 2: IDE892 Monotherapy Dose Expansion (MTAP-Deleted NSCLC) (Experimental): Participants with advanced or metastatic NSCLC with MTAP deletion will receive IDE892. One or more dose levels at or below the maximum tolerated dose from Part 1 will be further evaluated to determine the recommended Phase 2 dose and to assess antitumor activity.
  Interventions: Drug: IDE892
- Part 3: IDE892 + IDE397 Combination Dose Escalation (MTAP-Deleted Solid Tumors) (Experimental): Participants with advanced or metastatic solid tumors harboring MTAP deletion (including mesothelioma, gastroesophageal cancers, non-small cell lung cancer, and urothelial cancer) will receive IDE892 in combination with IDE397. Dose levels will be escalated using a modified toxicity probability interval (mTPI) design to evaluate safety, tolerability, and to determine the maximum tolerated dose and/or recommended dose for expansion. PK, PD, and preliminary antitumor activity will also be assessed.
  Interventions: Drug: IDE892; Drug: IDE397
- Part 4: IDE892 + IDE397 Combination Dose Expansion (MTAP-Deleted NSCLC) (Experimental): Participants with advanced or metastatic NSCLC with MTAP deletion will receive IDE892 in combination with IDE397. One or more dose levels at or below the maximum tolerated dose from Part 3 will be further evaluated to determine the recommended Phase 2 dose and to assess antitumor activity.
  Interventions: Drug: IDE892; Drug: IDE397

INTERVENTIONS:
Drug: IDE892 — IDE892 is an inhibitor of the Protein arginine methyltransferase 5 (PRMT5) that is being developed by IDEAYA Biosciences, Inc. as an anticancer therapeutic for patients with advanced or metastatic cancer harboring MTAP deletions.
Drug: IDE397 — IDE397 is an oral MAT2A inhibitor that is being developed by IDEAYA Biosciences, Inc. as an anticancer therapeutic for patients with advanced or metastatic cancer harboring MTAP deletions. In this study, IDE397 will be evaluated in combination with IDE892 (Parts 3 and 4) in participants with MTAP-deleted advanced solid tumors.
  Arms: Part 3: IDE892 + IDE397 Combination Dose Escalation (MTAP-Deleted Solid Tumors); Part 4: IDE892 + IDE397 Combination Dose Expansion (MTAP-Deleted NSCLC)

SUMMARY:
This is a multicenter clinical study to evaluate the safety, efficacy, and Pharmacokinetics (PK) of IDE892 as monotherapy and in combination with other agents including IDE397 in participants with methylthioadenosine phosphorylase (MTAP)-deleted advanced solid tumors within indications of interest.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate safety, efficacy, and PK of IDE892 as monotherapy and combination therapy in adult participants with MTAP-deleted tumors who have progressed after standard therapy and represent a high unmet need. In the current stage, the combination will be focused on IDE892 with IDE397, an oral inhibitor of methionine adenosyltransferase 2A (MAT2A), to fully exploit the vulnerabilities associated with methylthioadenosine (MTA) accumulation in MTAP-deleted tumors while maintaining a substantial therapeutic index. The mechanistic rationale for this study is discussed in the following sections.

ELIGIBILITY:
Inclusion Criteria:

* Are ≥ 18 years of age at the time of signing the ICF.
* Have a histologically confirmed diagnosis of a locally advanced recurrent or metastatic solid tumor type of interest with MTAP deletion (for dose escalation: mesothelioma [pleural or peritoneal], gastroesophageal cancers [squamous and adenocarcinoma of esophagus, gastric adenocarcinoma, gastroesophageal junction cancers], NSCLC [adenocarcinoma, squamous cell carcinoma, and adeno-squamous] and UC [including mixed urothelial-squamous histology]; for dose expansion: NSCLC that has progressed on at least one prior line of treatment and for which additional effective standard therapy is not available or for which the participant is not a candidate due to intolerance).
* Are willing and able to provide blood/tumor tissue samples for biomarker testing. An archival tumor tissue specimen must be provided for central confirmation of MTAP loss.
* Must be willing and able to provide the blood/serum/plasma samples
* Have evidence of homozygous loss of MTAP or MTAP deletion (pre-screening available after signing pre-screening ICF)
* Have at least 1 measurable lesion according to RECIST version 1.1
* Have Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 or 1
* Have life expectancy > 3 months
* Have adequate bone marrow and organ function
* Able to retain administered study drug/IMP.
* Male and female: willing to use contraception

Exclusion Criteria:

* Known symptomatic brain metastases requiring supraphysiologic doses of systemic corticosteroids
* Have a known primary central nervous system (CNS) malignancy
* Have had other malignancies within 2 years prior to the first dose, with some exceptions
* Impaired cardiac function or clinically significant cardiac diseases
* Have presence of uncontrolled pleural, peritoneal, or pericardial effusion within 2 weeks before the first study dose, requiring recurrent drainage procedures or an indwelling drainage catheter
* Have a history of severe infections within 4 weeks prior to the start of study treatment
* Hypertension (e.g., > 150/100 mmHg) that cannot be controlled by medications despite optimal medical therapy
* Other acute or chronic medical or psychiatric condition
* Have a history of immunodeficiency, with a positive human immunodeficiency virus(HIV) test at screening
* Known or suspected viral hepatitis
* Had an adverse reaction to a previous antitumor treatment that has not recovered to CTCAE Grade ≤ 1
* Have received chemotherapy within 3 weeks of the first dose of IMP; immunotherapy or biologic targeted antitumor treatments within 2 weeks before the first dose of IMP; small molecule inhibitors within 2 weeks before the first dose of IMP, or other investigational products within 4 weeks
* Current radiation-related toxicity or radiation therapy within 2 weeks before the first dose of IMP
* Administration of any of the following within 2 weeks before the first dose of IDE892 as a monotherapy: Strong inhibitors or inducers of cytochrome P450, Strong inhibitors of P-glycoprotein, Narrow therapeutic index and sensitive substrates of multidrug and toxin extrusion (MATE)1 and MATE2-K, Narrow therapeutic index and sensitive substrates of P-gp and breast cancer resistance protein
* Administration of any of the following within 2 weeks before the first dose of IDE892: Strong inhibitors or inducers of CYP3A4/5, Strong inhibitors of P-gp and/or BCRP, Narrow therapeutic index and sensitive substrates of MATE1 and MATE2-K, Narrow therapeutic index and sensitive substrates of P-gp and BCRP
* Use of proton pump inhibitors (PPIs) within 7 days prior to the first dose of IMP or planned use during the study
* Use of drugs with known risk for QT prolongation within 2 weeks prior to the first dose of IDE892
* Previous treatment with a MAT2A inhibitor and/or Protein arginine N-methyltransferase (PRMT) inhibitor
* Major surgery within 4 weeks before study entry
* Prior irradiation to > 25% of the bone marrow
* Known or suspected hypersensitivity to IDE892

Disease-Specific Eligibility Criteria NSCLC

* Must have histologically confirmed diagnosis of advanced or metastatic NSCLC that has progressed after prior treatment with platinum chemotherapy and a PD-1/PD-L1 inhibitor (unless contraindicated or participant developed intolerance) in the metastatic setting
* Treatment with no more than 3 prior lines, including no more than 2 prior lines of chemotherapy.
* If considered standard of care and available, participants whose cancers have proven targetable oncogene alterations must have had disease progression on (unless contraindicated or participant developed intolerance) at least 1 prior line containing appropriate targeted therapy.

Urothelial Cancer (Bladder and Upper Urinary Tract), Mesothelioma (Pleural or Peritoneal) and Gastroesophageal Cancers

* Must have histologically confirmed diagnosis of advanced or metastatic UC, mesothelioma, or gastroesophageal cancer
* Must have progressed following at least 1 prior line of therapy
* Treatment with no more than 3 prior lines, including no more than 2 prior lines of chemotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2026-02-28 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose-limiting Toxicities (DLTs) of IDE892 (Parts 1 and 3) | 21 days following the first dose of IDE892 (each cycle is 21 days)
  Incidence of DLTs of IDE892 will be determined in Parts 1 and 3
Incidence of AEs and SAEs (Parts 1, 2, 3, and 4) | From first dose until 28 days after last dose (each cycle is 21 days)
  Incidence and severity of adverse events (AEs)/serious adverse events (SAEs) (graded based on Common Terminology Criteria for Adverse Events [CTCAE] version 5.0) will be determined in Parts 1, 2, 3, and 4.
Objective response rate (ORR) and duration of response (DOR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 (Parts 2 and 4) | Approximately 2 years
  Objective response rate (ORR: best objective response of complete response [CR] + partial response [PR]) and duration of response (DOR) per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 as assessed by the Investigator

SECONDARY OUTCOMES:
Overall response rate (ORR) and duration of response (DOR) per RECIST version 1.1 (Parts 1 and 3) | Approximately 2 years
  ORR and DOR per RECIST version 1.1 as assessed by the Investigator
Disease control rate (DCR) and duration of stable disease per RECIST version 1.1 (Parts 1, 2, 3, and 4) | Approximately 2 years
  Disease control rate (disease control rate [DCR]: CR + PR + stable disease [SD]) and duration of SD per RECIST version 1.1 as assessed by the Investigator
Maximum Observed Plasma Concentration (Cmax) (Parts 1, 2, 3, and 4) | Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 21 days)
  Cmax is the highest observed plasma concentration of the study drug following administration of IDE892 as a single agent or in combination with IDE397
Time to Maximum Observed Concentration (Tmax) | Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 21 days)
  Time to Maximum Observed Concentration (Tmax) after administration of IDE892 as a single agent or in combination with IDE397
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUClast) | Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 21 days)
  AUClast reflects total drug exposure from dosing until the last measurable concentration after administration of IDE892 as a single agent or in combination with IDE397
Time of Last Quantifiable Concentration (Tlast) | Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 21 days)
  Tlast is the time at which the final measurable drug concentration is observed after administration of IDE892 as a single agent or in combination with IDE397
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUCinf) | Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 21 days)
  AUCinf represents total drug exposure extrapolated to infinite time after administration of IDE892 as a single agent or in combination with IDE397
Terminal Elimination Half-Life (t½) | Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 21 days)
  t½ is the time required for the plasma concentration of the drug to decrease by half during the terminal elimination phase after administration of IDE892 as a single agent or in combination with IDE397
Maximum Observed Plasma Concentration at Steady State (Cmax,ss) | Cycle 1 Day 15 (each cycle is 21 days)
  Cmax,ss is the maximum observed plasma concentration after achieving steady state after administration of IDE892 as a single agent or in combination with IDE397
Time to Maximum Concentration at Steady State (Tmax,ss) | Cycle 1 Day 15 (each cycle is 21 days)
  Tmax,ss is the time from dosing to Cmax at steady state after administration of IDE892 as a single agent or in combination with IDE397
Trough Plasma Concentration at Steady State (Ctrough) | Cycle 1 Day 15 (each cycle is 21 days)
  Ctrough is the concentration obtained immediately prior to the next scheduled dose at steady state after administration of IDE892 as a single agent or in combination with IDE397
Area Under the Plasma Concentration-Time Curve Over the Dosing Interval (AUCtau) | Cycle 1 Day 15 (each cycle is 21 days)
  AUCtau represents drug exposure over one full dosing interval at steady state after administration of IDE892 as a single agent or in combination with IDE397
Apparent Clearance (CL/F) | Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 21 days)
  CL/F is the apparent clearance of the drug after extravascular dosing after administration of IDE892 as a single agent or in combination with IDE397
Apparent Volume of Distribution (Vz/F) | Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 21 days)
  Vz/F is the apparent volume of distribution following extravascular dosing after administration of IDE892 as a single agent or in combination with IDE397
Accumulation Ratio (Rac) | Cycle 1 Day 1 and Cycle 1 Day 15 (each cycle is 21 days)
  Rac is calculated as the ratio of AUC or Cmax at steady state compared with first dose, reflecting drug accumulation after administration of IDE892 as a single agent or in combination with IDE397

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - NEXT Oncology Houston, Houston, Texas
  - NEXT Oncology Dallas, Irving, Texas
  - NEXT Oncology Virginia, Fairfax, Virginia